CLINICAL TRIAL: NCT04243538
Title: Developing and Piloting a Multi-component Technology-based Care Intervention to Address Patient Symptoms and Caregiver Burden in Home Hospice
Brief Title: Piloting a Multi-component Technology-based Care Intervention to Address Patient Symptoms in Home Hospice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Visiting Nurse Service of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-11022933frmrly19-04020138-1; 1K76AG059997-01A1 (NIH)
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Hospice

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Standard of care.
- I-HoME intervention (Experimental): Weekly televisits with a nurse practitioner that will implement the I-HoME intervention.
  Interventions: Behavioral: I-HoME

INTERVENTIONS:
Behavioral: I-HoME — I-HoME will consist of two components: (1) synchronous live video interactions between patients/CGs and a hospice nurse; and (2) educational videos.
  Arms: I-HoME intervention

SUMMARY:
With the growth of hospice, older adults have the opportunity to receive home-based care aimed at reducing suffering and focusing on quality of life at the end of life. While use of technology and educational videos has yet to be fully developed, structured, and evaluated in home hospice care, it has shown promise to improve care in other settings. Therefore, this study aims to develop and evaluate a multi-component technology-based care intervention, i.e., Improving Home hospice Management of End of life issues through technology (I-HoME).

DETAILED DESCRIPTION:
The study intervention focuses on assessing and addressing patient symptoms in the home hospice setting through weekly telehealth visits (for up to 6 weeks) and educational videos that are geared for the patient's informal caregiver. The aim of this phase of the project is two fold. One is that the study team will conduct a single armed (N=6 dyads) pilot study with a focus on optimizing data collection protocols and the intervention. After this step, a randomized pilot study evaluating the feasibility and potential efficacy of I-HoME (N=50 dyads) compared to usual care (N=50 dyads) will be conducted.

Phase I of the study to assess feasibility of the intervention was registered on ClinicalTrials.gov as NCT04074304.

ELIGIBILITY:
Inclusion Criteria:

Home hospice caregivers must be:

* English speaking
* 18 years of age or older
* not blind
* having a family member receiving home hospice care

Home hospice patients must be:

* English speaking
* 65 years of age or older
* not blind
* enrolled in home hospice care.

Exclusion Criteria:

* Patients with a terminal diagnosis of dementia or patients who have cognitive impairment and unable to sign a written informed consent will be excluded.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veerawat Phongtankuel, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The Visiting Nurse Service of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm | I-HoME Intervention
Started | 40 | 40
Completed | 40 | 35
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | I-HoME Intervention | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.91) | 60.6 (11.37) | 60.3 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 10 | 28
  Not Hispanic or Latino | 22 | 30 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 11 | 23
  White | 17 | 17 | 34
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Highest Education Completed [Count of Participants; unit: Participants]
  Some high school | 2 | 1 | 3
  High School or GED | 4 | 3 | 7
  Some College | 10 | 11 | 21
  College degree | 10 | 9 | 19
  Post-graduate but no degree | 2 | 2 | 4
  Graduate Degree | 12 | 14 | 26
Relationship to Patient [Count of Participants; unit: Participants]
  Spouse/partner | 6 | 8 | 14
  Child | 28 | 26 | 54
  Relative | 5 | 6 | 11
  Friend | 1 | 0 | 1
Annual Household Income Range [Count of Participants; unit: Participants]
  $25,000 or less | 8 | 3 | 11
  $25,001 to $50,000 | 11 | 11 | 22
  $50,001 to $75,000 | 8 | 10 | 18
  $75,001 or greater | 13 | 15 | 28
  Declined to answer | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participant Recruitment Rate
Description: Recruitment rate was measured by the number of participants consented divided by the number of eligible participants.
Time Frame: During recruitment (22 months)
Population: All participants who we reached out to and were eligible for our study, including those who refused to participate, were unreachable over multiple attempts, and those who were initially interested in participating but not enrolled were included in the number of participants analyzed for this measure.
Measure: Number; unit: percentage of enrolled participants
Groups:
- All Participants: This measure represents the recruitment rate for all participants.
Arm/Group | All Participants
Number analyzed (Participants) | 212
percentage of enrolled participants | 37.7

2. Primary Outcome: Participant Attrition From Enrollment to End of Study
Description: This measure is the total number of participants who withdrew consent or were unreachable for study activities after consent.
Time Frame: At the end of the intervention or at 6 weeks, which ever is earlier.
Population: This measure includes all participants who were enrolled.
Measure: Count of Participants; unit: Participants
Groups:
- I-HoME Intervention: I-HoME consists of two components: (1) a weekly tele-visit with a hospice nurse practitioner for up to 6 weeks, and (2) caregiver educational videos.
Arm/Group | Control Arm | I-HoME Intervention
Number analyzed (Participants) | 40 | 40
Participants | 0 | 5

3. Primary Outcome: Average Length of I-HoME Tele-visit
Description: This measure was collected by calculating the average duration (in minutes) of each tele-visit between the participant in I-HoME intervention arm and the interventionalist.
Time Frame: At the end of the intervention or at 6 weeks, which ever is earlier.
Population: The measure was only assessed for the intervention arm. 5 subjects were excluded for this measure because 2 participants withdrew consent and 3 participants were lost to follow up, thus not receiving the intervention.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Arm | I-HoME Intervention
Number analyzed (Participants) | 0 | 35
minutes |  | 22.5 (11.32)

4. Primary Outcome: Total Number of Educational Videos Watched by I-HoME Intervention Arm Participants
Description: This measure is the total number of videos watched by the I-HoME intervention arm participants who received at least one tele-visit. Intervention arm participants self-reported whether they watched the educational videos recommended to them by the interventionist.
Time Frame: At the end of the intervention or at 6 weeks, which ever is earlier.
Population: as for outcome 3
Measure: Number; unit: videos
Arm/Group | Control Arm | I-HoME Intervention
Number analyzed (Participants) | 0 | 35
videos |  | 23

5. Primary Outcome: Number of I-HoME Intervention Caregivers Who Experienced Technical Issues During the Tele-visits.
Description: The number of I-HoME intervention caregivers who reported at least one technical issues with the tele-visit. Participants in the intervention arm answered questions about whether they experienced technical issues.
Time Frame: At the end of the intervention or at 6 weeks, which ever is earlier.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | I-HoME Intervention
Number analyzed (Participants) | 0 | 35
Participants
  Reported Technical Issues | 0 | 13
  Did Not Report Technical Issues | 0 | 22

6. Primary Outcome: Percentage of Tele-visits With Hardware Issues Out of the Total Number of Tele-visit Intervention Visits
Description: After each intervention visit, participants answered questions about whether they experienced technical issues. This measure was calculated by dividing the number of I-HoME tele-visits during which the participant and/or the interventionist experienced hardware issues by the total number of I-HoME tele-visits administered during the entire study period.
Time Frame: At the end of the intervention or at 6 weeks, which ever is earlier.
Population: This measure was unable to be collected because it was difficult to distinguish hardware issues from other technical issues, which were reported in Primary Outcome #5.
Arm/Group | Control Arm | I-HoME Intervention
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Percentage of Tele-visits Conducted Out of the Total Possible Tele-visits.
Description: This measure is calculated by dividing the tele-visits conducted out of the total possible tele-visits. This measure shows the adherence of the I-HoME intervention arm to the tele-visits.
Time Frame: At the end of the intervention or at 6 weeks, which ever is earlier.
Population: The total number of tele-visits completed by the I-HoME intervention arm participants was divided by the intended number of tele-visits for this group. The measure was only assessed for the intervention arm. 5 subjects were excluded for this measure because 2 participants withdrew consent and 3 participants were lost to follow up, thus not receiving the intervention.
Measure: Number; unit: percentage of tele-visits conducted out
Arm/Group | Control Arm | I-HoME Intervention
Number analyzed (Participants) | 0 | 35
percentage of tele-visits conducted out |  | 89.6

8. Secondary Outcome: Patients' Symptom Burden Score as Rated by the Caregiver, Measured at Baseline and Weekly for 6 Weeks.
Description: Symptom burden score as measured by the Edmonton Symptom Assessment Scale (ESAS). Scale is from a 0 to 90, with higher scores indicating higher symptom burden.
Time Frame: At baseline and weekly for 6 weeks.
Population: This analysis included participants who completed the six-week study. The number of participants analyzed at each time point varied because:
  1. Caregiver attrition
  2. The caregiver did not answer one or more questions on the survey
  3. The caregiver was ineligible to participate due to their care recipient passing away or being discharged from hospice
  4. Caregivers in the intervention arm missed the tele-visit session on that particular week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | I-HoME Intervention
Number analyzed (Participants) | 34 | 17
score on a scale
  Baseline ESAS Score: number analyzed (Participants) | 33 | 15
  Baseline ESAS Score | 39.0 (13.9) | 43.7 (17.6)
  Week 1 ESAS Score: number analyzed (Participants) | 30 | 14
  Week 1 ESAS Score | 38.0 (16.7) | 40.7 (19.6)
  Week 2 ESAS Score: number analyzed (Participants) | 29 | 13
  Week 2 ESAS Score | 34.6 (15.1) | 42.5 (16.8)
  Week 3 ESAS Score: number analyzed (Participants) | 33 | 11
  Week 3 ESAS Score | 34.7 (15.9) | 42.3 (16.1)
  Week 4 ESAS Score: number analyzed (Participants) | 31 | 12
  Week 4 ESAS Score | 34.9 (16.5) | 38.8 (19.2)
  Week 5 ESAS Score: number analyzed (Participants) | 28 | 14
  Week 5 ESAS Score | 37.0 (16.1) | 44.1 (17.9)
  Week 6 ESAS Score: number analyzed (Participants) | 33 | 14
  Week 6 ESAS Score | 36.1 (15.6) | 39.9 (20.1)

9. Secondary Outcome: Number of Patient Hospitalizations From Enrollment to End of Intervention
Description: All hospitalizations of the caregivers' patient from enrollment to end of intervention
Time Frame: From enrollment to the end of the intervention or at 6 weeks, which ever is earlier.
Population: This data was unable to be collected because we didn't have access to the patients' medical records after they were discharged to accurately determine whether they were hospitalized after hospice discharge.
Arm/Group | Control Arm | I-HoME Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Control Arm | I-HoME Intervention
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT04243538/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT04243538/ICF_001.pdf